CLINICAL TRIAL: NCT02070224
Title: Evaluation of the Prognostic Value of Biological Markers, Coll2-1 and Coll2-1NO2 in Patients With Symptomatic Knee Osteoarthritis
Acronym: PRODIGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Artialis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PRODIGE
Record Dates: First submitted 2014-02-19; First posted 2014-02-25 (Estimated); Last update posted 2019-02-05 (Actual); Status verified 2017-01

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — X-Rays; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Knee osteoarthritis (Other)
  Interventions: Other: Serum and urine samples collections; Other: Imaging (x-rays and MRI)

INTERVENTIONS:
Other: Serum and urine samples collections — Serum and urine samples will be collected at baseline, 3 month, 6 month, 12 month to assess the predictive value of cartilage-specific biomarkers Coll2-1/Coll2-1NO2 on OA progression (MRI, Clinical and radiological progression)
Other: Imaging (x-rays and MRI) — MRI will be done at baseline and 12 month and x-rays will be done at baseline

SUMMARY:
The purposes of this study are to assess the prognostic value of serum and urinary biomarkers Coll2-1 and Coll2-1NO2 at baseline, and their change over the first year, on the progression of knee osteoarthritis MRI scores at 12 months, on the progression of knee osteoarthritis clinical score at 12 months. Additionally, this study will search for correlations between serum and urinary biomarkers Coll2-1 and Coll2-1NO2 at baseline with the radiographic, MRI and clinical severity of knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 45 to 80 years with a BMI ≤ 40
* With an uni- or bilateral femorotibial knee osteoarthritis associated or not with a femoro-patellar knee osteoarthritis
* Responding to clinical and radiological criteria of the ACR
* Symptomatic for more than 6 months (for the most painful knee)
* K&L radiological grade of Felson II or III
* With a cartilage lesion identified during MRI and either at least 1 out of 4 MRI severity criteria:

  * bone oedema
  * meniscal lesion in the central region of the medial compartment
  * effusion without answer to corticosteroids
  * zone without cartilage
* or at least 1 out of 3 clinical severity criteria:

  * genu varum>3°
  * previous meniscal surgery
  * known polyarthritis
  * effusion on the target knee
* Sign an informed consent after being informed
* Able to follow the instructions of the study
* With an agreement from the physicians having established the diagnosis of osteoarthritis (if any) to give relevant information to the investigator
* With health insurance (for France).

Exclusion Criteria:

For osteoarthritis:

* Isolated patellofemoral arthritis
* Chondromatosis or villo-nodular synovioma of the knee
* Recent trauma-induced knee pain
* Joint disease due to joint dysplasia, aseptic osteonecrosis, acromegaly, Paget's disease, hemophilia, hemochromatosis, …
* inflammatory pathologies as rheumatoid polyarthritis, gout arthritis, infectious arthritis
* Diseases that may interfere with the evaluation of osteoarthritis (radiculalgia of lower limbs, arteritis, …)
* Genu valgum (degree considered as pathological by the physician)

For previous treatments:

• Treatment with strontium ranelate, bisphosphonates, SERM and PTH

For known associated diseases:

* Serious associated diseases: severe liver or renal failure, uncontrolled cardiovascular disease, HIV, hepatitis B or C
* Knee tumor

For patients:

* Patient who participated to a therapeutic clinical trial 3 months before the T0 inclusion visit
* Patient who are the subject of a judicial protection measure or under guardianship
* Pregnant woman

For MRI contraindications:

* Patient with a pacemaker, an implantable defibrillator, neurosurgical clips, a neurostimulator, cochlear implant, a stent, an insulin pump
* Patient with a ferromagnetic splinter in the body, or having wire sutures
* Serious mobility problem (Parkinson, tremors)

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-01; Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
MRI will be analysed with semiquantitative Whole-Organ Magnetic Resonance Imaging Scoring method (WORMS) | 12 month

SECONDARY OUTCOMES:
Knee injury and Osteoarthritis Outcome Score (KOOS) and Visual Analogue Scales (VAS) for mean knee pain and global patient assessment of disease activity | 12 month

OTHER OUTCOMES:
Knee prosthesis during the study | 12 month
MRI cartilage volume (optional) | 12 month
MRI T2 relaxation time (optional) | 12 month
MRI MOAKS scoring (optional) | 12 month

CONTACTS AND LOCATIONS:
Locations (2):
- University Hospital of Liege-CHU, Liège, Belgium
- University Hospital of Nancy, Nancy, France

REFERENCES:
- [Derived] Hick AC, Malaise M, Loeuille D, Conrozier T, Maugars Y, Pelousse F, Tits C, Henrotin Y. Cartilage Biomarkers Coll2-1 and Coll2-1NO2 Are Associated with Knee OA MRI Features and Are Helpful in Identifying Patients at Risk of Disease Worsening. Cartilage. 2021 Dec;13(1_suppl):1637S-1647S. doi: 10.1177/19476035211021892. Epub 2021 Jun 15. PMID 34128409
- [Derived] Hick AC, Fonck M, Costes B, Cobraiville E, Pirson S, Garcia L, Labasse A, Vander Poelen S, Henrotin Y. Serum Levels of Coll2-1, a Specific Biomarker of Cartilage Degradation, Are Not Affected by Sampling Conditions, Circadian Rhythm, and Seasonality. Cartilage. 2021 Dec;13(1_suppl):540S-549S. doi: 10.1177/1947603519878489. Epub 2019 Oct 20. PMID 31631693